CLINICAL TRIAL: NCT05815095
Title: Randomized Pragmatic, Cluster, Stepped-wedge Trial of Early Detection and Referral for Autism and Neurodevelopmental Disorders at the Maternal and Child Protection Services for Care Before 1 Year of Follow-up
Brief Title: Early Detection and Referral for Autism and Neurodevelopmental Disorders at the Maternal and Child Protection Services
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PRECO TSA
Record Dates: First submitted 2023-03-09; First posted 2023-04-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: Autism Spectrum Disorder / diagnosis; Neurodevelopmental Disorders /diagnosis; Infant; Prospective Study
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine practice (control): In this group, a health professional will assess the infant's neurodevelopmental characteristics through routine practice evaluations, such as motor skills, vocalizations, babbling, and social interactions
- Use of PREAUT Grid (intervention): In this group, a health professional will assess the infant's neurodevelopmental characteristics using the PREAUT grid
  Interventions: Other: PREAUT grid

INTERVENTIONS:
Other: PREAUT grid — Patient with abnormal results in this evaluation would be referred to a specialized center early for advice and treatment if necessary
  Groups: Use of PREAUT Grid (intervention)

SUMMARY:
This study aims to compare two screening strategies for identifying infants with a potential risk of Autism Spectrum and Neurodevelopmental Disorders to provide early access to care and increase the likelihood of a favorable outcome

DETAILED DESCRIPTION:
This prospective cohort study is performed at several Maternal and Child Protection Services in France. It aims to early detect infants under 12 months of age with a developmental gap compared to that expected for their age.

The first consultation will occur at the same time as the infant's usual medical follow-up at the Maternal and Child Protection Service (usually vaccination in the fourth month and developmental examination at nine months). Two strategies will be evaluated during this visit to assess the infant's neurodevelopmental characteristics. In the first one, a health professional will assess the infant's neurodevelopmental characteristics through routine practice evaluations, such as motor skills, vocalizations, babbling, and social interactions. In the second one, the PREAUT grid will be used for screening of screening for autism spectrum disorder.

Patients with abnormal results in these evaluations would be referred to a specialized center early for advice and treatment if necessary. We will consider an early referral as the referral of infants to an adapted consultation within the month following the first consultation. Also, these patients will be assessed using the State-Trait Anxiety Inventory-Form Y and T and the QUALIN score.

After 12 months of follow-up, data regarding the received treatments of patients who were addressed to a specialized center will be performed.

At 24 and 36 months of follow-up, all the included patients will be assessed with the Modified Checklist for Autism in Toddlers, Revised with Follow-up instrument (M-CHAT-R/F) ,and the IDE ( the French version of the Child Development Inventory). In case of an abnormal result of the M-CHAT-R/F, the Autism Diagnostic Interview-Revised (ADI-R) and the Autism Diagnostic Observation Schedule (ADOS) will be administered. In case of an abnormal result of the IDE, the Brunet-Lézine scale will be administered.

Finally, the French health insurance claims databases will be used to evaluate the care pathway of all included patients up to 48 months of the child.

ELIGIBILITY:
Inclusion Criteria:in

* Infants between 4 and 9 months of age followed up in the participating Maternal and Child Protection Services for the fourth and ninth-month mandatory vaccinations
* Availability of a personnel telephone for at least one parent
* Information to the parents for data collection and the active follow-up of the child until 36 months and express consent to participate in the research
* Affiliation to a social security system or benefiting from the Medical assistance of the state
* Mastery of a minimum of French according to the principal investigator or the presence of a French-speaking relative

Exclusion Criteria:

* Infant with a severe neurological pathology such as encephalopathy
* Refusal to participate in the study

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged at least 4 months at study inclusion and followed in Maternal and Child Protection Services
Sampling Method: Non-Probability Sample
Enrollment: 10400 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2030-04-14 (Estimated); Study Completion 2032-04-14 (Estimated)

PRIMARY OUTCOMES:
Proportion of children at 24 months with an Autism Spectrum Disorder or Neurodevelopmental Disorder diagnosis who received care before the age of one | At 2 years of age

SECONDARY OUTCOMES:
Effectiveness of two screening strategies on the occurrence severity of Autism Spectrum Disorders (ASD) and Neurodevelopmental Disorders (NDD) | At 2 and 3 years of age
Predictive performance of the PREAUT grid (at four months and nine months) compared to the usual diagnosis | At 2 and 3 years of age
Association between ASD-NDD diagnosis and neonatal or familial risk factors | At 2 and 3 years of age of child's referral to the Medical psychological center
Quality of life assessed by the QUALIN score | At inclusion in Maternal and Child Protection Services or at Medical-psychological center and at 2 and 3 years of age
Measurement of the parents' psychological state at the time of the child's referral to the Medical psychological center | At a Medical-psychological center and at 2 and 3 years of age
Impact on the family life (IOFS) of a child diagnosed with risk of Autism Spectrum and Neurodevelopmental Disorders | At 2 and 3 years of age
Evaluation of the implementation of the new model of systematic screening of infants in Maternal and Child Protection Services and systematic referral to the Medical-psychological center | Through study completion, an average of 4 years
Evaluation of the implementation of infant care in the Medical-psychological center | Through study completion, an average of 4 years
Qualitative study of the incentives and obstacles of the screening and early referral strategy with the Maternal and Child Protection Service's workers | Through study completion, an average of 4 years
Qualitative study of the screening and early referral strategy with parents | Through study completion, an average of 4 years
Description of the practice of identification by the Maternal and Child Protection Services and referral to the Medical-psychological center | At the inclusion, at the end of inclusion and at the late visit
Description of the care pathway in the two groups | At 4 years of the child

CONTACTS AND LOCATIONS:
Locations (1):
- PMI Stalingrad, Champigny-sur-Marne, France

REFERENCES:
- [Derived] Delmas C, Wang XX, Pelloux AS, Caeymaex L, Bouaziz N, Aegerter P, Jung C. Effectiveness of early detection and coordinated referral of infants before 1 year at risk for autism spectrum and neurodevelopmental disorders in maternal and child protection centre: a French randomised pragmatic trial in a stepped-wedge trial (PRECO-TSA protocol). BMJ Open. 2025 Aug 4;15(8):e094729. doi: 10.1136/bmjopen-2024-094729. PMID 40759525